CLINICAL TRIAL: NCT04472221
Title: Arterio-arterial Vascular Access as a Novel Technique for Treatment of Venous Hypertention With Arterio-venous Vascular Access
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R.20.06.909 - 2020/06/24
Record Dates: First submitted 2020-07-01; First posted 2020-07-15 (Actual); Last update posted 2020-07-15 (Actual); Status verified 2020-07

CONDITIONS: Vascular Access Complication

STUDY DESIGN:
Intervention Model Description: Experimental
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vascular Access Venous Hypertension (Experimental): Swollen upper limb with synthetic Arteriovenous graft
  Interventions: Procedure: Arterioarterial synthetic graft

INTERVENTIONS:
Procedure: Arterioarterial synthetic graft — Synthetic poly tetraflouroethylene graft

SUMMARY:
Arterio-arterial vascular access, Arterio-venous synthetic access, Venous hypertension, Hemodialysis patients Purpose: To describe a technique used to treat a patient with Lt upper limb synthetic arterio-venous vascular access and venous hypertension of the same limb. Technique: the investigator expose the venous anastomosis of the graft by small longitudinal incision in the axilla and dissection of the axillary artery just parallel to the axillary vein , the investigator disconnect the graft from the axillary vein and do primary repair of the vein , then the investigator do end to side anastomosis of the graft to the axillary artery , after finishing this anastomosis the axillary artery ligated just below the anastomosis. Conclusion: the conversion of arterio-venous graft to arterio-arterial vascular access in precious access with venous hypertension lead to resolution of edema of venous hypertension and preservation of access for dialysis.

DETAILED DESCRIPTION:
Abstract Purpose: To describe a technique used to treat a patient with Lt upper limb synthetic arterio-venous vascular access and venous hypertension of the same limb. Technique: we expose the venous anastomosis of the graft by small longitudinal incision in the axilla and dissection of the axillary artery just parallel to the axillary vein , the investigator disconnect the graft from the axillary vein and do primary repair of the vein , then investigator s do end to side anastomosis of the graft to the axillary artery , after finishing this anastomosis the axillary artery ligated just below the anastomosis. Conclusion: the conversion of arterio-venous graft to arterio-arterial vascular access in precious access with venous hypertension lead to resolution of edema of venous hypertension and preservation of access for dialysis.

Keywords: Arterio-arterial vascular access, Arterio-venous synthetic access, Venous hypertension, Hemodialysis patients.

Introduction:

In haemodialysis patients the investigator are confronted by patient with Left upper limb synthetic graft used for haemodialysis and the patient developed edema due to central venous occlusion ( venous hypertension) in the same limb. The other limb have no palpable pulse due to previous 3 operations for vascular access which ended by ligation of the brachial artery.

First the hope to dilatation of the central veins but this trial failed due to failure of the wire to cross the lesion, so we think to convert this arterio-venous graft to arterio-arterial access as we have previous experience with brachial aretrio-arterial vascular access.

One limitation of this technique was that the continuity of the brachial artery which will lead to thrombosis of the graft because of equal pressure in the graft and the brachial artery so ligation of the axillary artery below the proximal anastomosis was done despite our fear of ischaemia of the limb if the synthetic graft occluded later on.

Technique:

After failure of trial angioplasty of epsilateral central veins. This procedure was done either by local, regional, or general anesthesia (IV deprivan) according to the patient situation and surgeon preference.

Longitudinal incision (about 5-7cm) in the axilla at the arterio-venous anastomosis of the synthetic graft and along the course of the axillary artery , good hemostasis is needed because of the edema and the venous hypertension in the dilated collateral veins.

Good exposure of the end of the synthetic graft and mobilization of the axillary artery was done with ligation of intervening branches (a segment of 4-6 cm).

The synthetic graft catted and we do repair of the axillary vein. End to side anastomosis between the synthetic graft and the axillary artery by 6/0 proline then the axillary artery is ligated just below the anastomosis by 2/0 silk suture , now the blood is reversed in the synthetic graft and the blood flow from the axillary artery to the synthetic graft then to the brachial artery and radial and ulnar arteries.

Patients were discharged in the 2nd postoperative day unless need. Creep bandage was applied to the forearm and after 1-2 days the edema resolved and the patient regain the function of the upper limb and he can used the graft for dialysis immediately because the graft already healed and used previously for dialysis which is useful in those patients who has no venous access even for temporary catheter .

The same instructions as any arterio-arterial graft for hemodialysis were given to the patient and the medical stuff at dialysis unit as:

* no medications given at the AAPL to avoid intra-arterial injection and acute ischemia.
* Only pulse which can be palpated at the graft but no thrill.
* Patency of the graft is done by palpation of the distal pulsation (distal brachial or radial artery) or duplex.
* The puncture site needs more time of compression than that needed for AV grafts. (Khafagy et al.,)

ELIGIBILITY:
Inclusion Criteria:

* All vascular access with central venous hypertension with failed angioplasty

Exclusion Criteria:

* infected access or rupture access

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-06-21 (Actual); Primary Completion 2021-06-21 (Estimated); Study Completion 2021-06-21 (Estimated)

PRIMARY OUTCOMES:
Decrease the swelling of the upper limb gradually | Six month
  Measure of the whole cicumference
Patency of the dialysis access | Six month
  Duplex ultrasound assessment of the patency
Effeicient dialysis | 4 hours
  Continue haemodialysis of the access for 4 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura University, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No